CLINICAL TRIAL: NCT00479375
Title: Randomized Controlled Trial of Human Papillomavirus Testing in Primary Cervical Screening
Brief Title: Randomized Controlled Trial of Human Papillomavirus Testing in Primary Cervical Cancer Screening
Acronym: SWEDESCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Swedish Cancer Society (Other); Europe Against Cancer (European Union Directorate General XII- Public Health) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 3824-B00-05XAC
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia
Keywords: screening; human papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Adding Human Papillomavirus testing to organised cervical screening

SUMMARY:
Human papillomavirus (HPV)-based cervical screening is known to increase sensitivity for detection of high-grade cervical intraepithelial neoplasia (CIN). Randomized trials of longitudinal efficacy are required to assess whether these gains represent overdiagnosis or a protective effect.

Methods: A total of 12527 women, aged 32-38, attending population-based invitational screening in Sweden were randomized 1:1 to HPV test and cytology (intervention arm) or cytology only (control arm). HPV-positive women were invited for a second HPV test at least one year later and women with type-specific persistent infections were then invited to colposcopy. A similar number of random double-blinded procedures are performed in the control arm. Women are followed with comprehensive registry-based follow-up. Primary outcome is the relative rates of CIN grade 2 or worse (CIN2/CIN3+) found in subsequent screening. Secondary outcomes are the relative rates of CIN2/CIN3+ found in the aseline screening and outcomes stratified by grade of CIN (CIN 2 or CIN3+).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 32-38 years old
* Attending the Swedish population-based organised cervical screening program

Exclusion Criteria:

* Not providing informed consent

Ages: 32 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12527 (Actual)
Dates: Start 1997-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Incidence of CIN2/CIN3+ lesions (which includes invasive cancers and in situ adenocarcinomas) found by subsequent screening (i.e. after the enrollment screening round and its associated follow-up). | On average 4 years post baseline

SECONDARY OUTCOMES:
Secondary outcomes were the incidence of CIN2/CIN3+ lesions at enrollment screening (including associated follow-up) and outcomes stratified by CIN2 and CIN3+ lesions as endpoints. | On average 4 years post baseline
Re-analysis of primary and secondary outcomes also after subsequent 3-yearly screening rounds | On average 7, 10, 13 (et cetera) years post base-line

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD, Principal Investigator — Malmo University Hospital, Lund University
Locations (1):
- Malmo University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Forslund O, Antonsson A, Edlund K, van den Brule AJ, Hansson BG, Meijer CJ, Ryd W, Rylander E, Strand A, Wadell G, Dillner J, Johansson B. Population-based type-specific prevalence of high-risk human papillomavirus infection in middle-aged Swedish women. J Med Virol. 2002 Apr;66(4):535-41. doi: 10.1002/jmv.2178. PMID 11857534
- [Result] Elfgren K, Rylander E, Radberg T, Strander B, Strand A, Paajanen K, Sjoberg I, Ryd W, Silins I, Dillner J; Swedescreen Study Group. Colposcopic and histopathologic evaluation of women participating in population-based screening for human papillomavirus deoxyribonucleic acid persistence. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):650-7. doi: 10.1016/j.ajog.2005.01.056. PMID 16150255
- [Derived] Wang J, Elfstrom KM, Lagheden C, Eklund C, Sundstrom K, Sparen P, Dillner J. Impact of cervical screening by human papillomavirus genotype: Population-based estimations. PLoS Med. 2023 Oct 27;20(10):e1004304. doi: 10.1371/journal.pmed.1004304. eCollection 2023 Oct. PMID 37889928
- [Derived] Elfstrom KM, Smelov V, Johansson AL, Eklund C, Naucler P, Arnheim-Dahlstrom L, Dillner J. Long term duration of protective effect for HPV negative women: follow-up of primary HPV screening randomised controlled trial. BMJ. 2014 Jan 16;348:g130. doi: 10.1136/bmj.g130. PMID 24435414
- [Derived] Naucler P, Ryd W, Tornberg S, Strand A, Wadell G, Elfgren K, Radberg T, Strander B, Johansson B, Forslund O, Hansson BG, Rylander E, Dillner J. Human papillomavirus and Papanicolaou tests to screen for cervical cancer. N Engl J Med. 2007 Oct 18;357(16):1589-97. doi: 10.1056/NEJMoa073204. PMID 17942872